CLINICAL TRIAL: NCT05255770
Title: A Double Masked, Randomised, 3-way Cross-over, Single-center, Clinical Investigation to Evaluate the Effectiveness of Two NRL Condoms With Benzocaine Paste Compared With a Standard NRL Control in Prolonging Time to Ejaculation in Healthy Adult Men
Brief Title: A Clinical Investigation to Assess the Effectiveness of Benzocaine Condoms in Healthy Adult Men
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of the product development strategy
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 5061901
Record Dates: First submitted 2021-12-23; First posted 2022-02-25 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Ejaculation Delayed
MeSH Terms: conditions — Ejaculatory Dysfunction

STUDY DESIGN:
Intervention Model Description: The condom types will be tested in a 3-way cross-over design where subjects will be randomised to use each of the 3 condom types in a defined order, according to the randomisation schedule.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Each condom will be contained within an individual foil packet on which all branding will be masked. All the condom types will be masked in the same manner and identical secondary packaging boxes will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test condom A (NRL condom with 5% benzocaine paste) (Experimental): Following randomisation each subject will be given one set of 8 condoms as per randomisation schedule. After reporting at least 4 duration records (from vaginal entry to ejaculation), subjects will return to the clinical site for collection of their next set of condoms.
  Interventions: Device: Test condom A (NRL condom with 5% benzocaine paste); Device: Test condom B (NRL condom with 3% benzocaine paste); Device: Control NRL condom
- Test condom B (NRL condom with 3% benzocaine paste) (Experimental): Following randomisation each subject will be given one set of 8 condoms as per randomisation schedule. After reporting at least 4 duration records (from vaginal entry to ejaculation), subjects will return to the clinical site for collection of their next set of condoms.
  Interventions: Device: Test condom A (NRL condom with 5% benzocaine paste); Device: Test condom B (NRL condom with 3% benzocaine paste); Device: Control NRL condom
- Control NRL condom (Active Comparator): Following randomisation each subject will be given one set of 8 condoms as per randomisation schedule. After reporting at least 4 duration records (from vaginal entry to ejaculation), subjects will return to the clinical site for collection of their next set of condoms.
  Interventions: Device: Test condom A (NRL condom with 5% benzocaine paste); Device: Test condom B (NRL condom with 3% benzocaine paste); Device: Control NRL condom

INTERVENTIONS:
Device: Test condom A (NRL condom with 5% benzocaine paste) — In each assessment period (intervention duration), subjects will be provided with a condom type to use during vaginal intercourse and will report at least 4 duration records (from vaginal entry to ejaculation) over a 4-week period.
Device: Test condom B (NRL condom with 3% benzocaine paste) — In each assessment period (intervention duration), subjects will be provided with a condom type to use during vaginal intercourse and will report at least 4 duration records (from vaginal entry to ejaculation) over a 4-week period.
Device: Control NRL condom — In each assessment period (intervention duration), subjects will be provided with a condom type to use during vaginal intercourse and will report at least 4 duration records (from vaginal entry to ejaculation) over a 4-week period.

SUMMARY:
This investigation is designed to evaluate the effectiveness of two NRL condoms with Benzocaine paste compared with a standard NRL control.

DETAILED DESCRIPTION:
In this clinical investigation, two NRL condoms with Benzocaine paste (Test condom A and Test condom B) will be evaluated against a standard NRL male condom (Control condom) in prolonging time to ejaculation in healthy adult men.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects and their female partners between the ages of >=18 years and =<60 years.
2. Subjects and their female partners must have no health condition in their medical history.
3. Subject must be sexually active having regular intercourse (a minimum frequency of once a week).
4. Subjects in a stable, monogamous, sexual relationship with the same female partner for more than or equal to 3 months.
5. Subject's female partner should already be on an established other highly effective form of non-barrier contraception, unless post-menopausal.

Exclusion Criteria:

1. Subject or his female partner with alcohol or drug abuse.
2. Subjects and their female partners with anemia, coronary artery disease, impaired cardiac conduction, pulmonary disease, diabetes, and renal or hepatic disease.
3. Subjects and their female partners with a risk of methaemoglobinemia / complications related to ester anaesthetics which could trigger methemoglobinemia.
4. Subject and/or his female partner with urological disease or genitourinary surgery; ongoing significant psychiatric disorder not controlled by medication; history of surgery or injury to the pelvis, retroperitoneal surgery, radiotherapy, multiple sclerosis, spinal cord injury, chronic inflammation of the prostate or urethra; relevant genital surgery; a female partner with vaginal complaints; any broken skin or wounds in the genital area.
5. Subjects on medication that is contraindicated, which may affect erection.
6. Subject and/or his female partner have any medication which may affect the safety of the subject, including but not limited to benzocaine drug interactions such as Sulphonamides and cholinesterase inhibitors.
7. Subject with premature ejaculation, erectile dysfunction, hypo or hyperthyroidism, hypogonadism, hyperprolactinemia, ejaculatory dysfunction, haemorrhagic disorder, hepatitis B or C, human immunodeficiency virus (HIV) infection or having had penile implant surgery.
8. Subjects and their female partners who have any relevant history of allergy including local anaesthetics, parabens, PABA, commercial hair dyes, paraphenylenediamine, lubricants and latex.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male subjects who will use male condoms for intravaginal intercourse.
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
To determine the effectiveness of the Test Condom A compared with the Control NRL Condom at prolonging time to ejaculation. | 4 weeks for each assessment period (intervention duration)
  Subjects will be recording the duration (time in minutes:seconds) from vaginal entry to ejaculation for each condom use. The outcome is evaluated by the change from baseline with the Test Condom A compared to the Control NRL Condom, over a 4-week assessment period.

SECONDARY OUTCOMES:
To determine the effectiveness of the Test Condom B compared with the Control NRL Condom at prolonging time to ejaculation. | 4 weeks for each assessment period (intervention duration)
  Subjects will be recording the duration (time in minutes:seconds) from vaginal entry to ejaculation for each condom use. The outcome is evaluated by the change from baseline with the Test Condom B compared to the Control NRL Condom, over a 4-week assessment period.
To determine the effectiveness of the Test Condom A and Test Condom B compared with the Control NRL Condom at prolonging time to ejaculation for an increase of 2, 3, and 4 minutes. | 4 weeks for each assessment period (intervention duration)
  Subjects will be recording the duration (time in minutes:seconds) from vaginal entry to ejaculation for each condom use. The outcome is evaluated by the proportion of subjects who achieve an increase of 2, 3 and 4 minutes from baseline in each of the Test Condom A and Test Condom B compared to the Control NRL Condom.
To evaluate the sexual pleasure when using the Test Condom A or Test Condom B compared with the Control NRL Condom. | 4 weeks for each assessment period (intervention duration)
  The outcome is assessed by the measure of EMSEX (Event-level Male Sexual) pleasure scale questionnaire, a subject perceived questionnaire, at the end of a 4-week assessment period when using Test Condom A or Test Condom B compared with the Control NRL Condom.
To evaluate the subject's improvement at "lasting longer" for both the Test Condom A and Test Condom B compared with the Control NRL Condom. | 4 weeks for each assessment period (intervention duration)
  The outcome is assessed by the measure of Patient Global Impression of Change (PGIC), a subject perceived questionnaire, at the end of a 4-week assessment period when using Test Condom A or Test Condom B compared with the Control NRL Condom.
Subject's experience on the use of each type of condoms [Acceptability and In-Use Tolerability] | 19 weeks
  Acceptability and in-use tolerability as assessed by subject perceived questionnaires.

IPD SHARING:
Plan to Share IPD: No
IPD will be shared as per local regulations.